CLINICAL TRIAL: NCT00573716
Title: A Comparison of Bone Mineral Density Changes During Treatment With Risperidone or Aripiprazole in Adolescents
Brief Title: Comparison of Bone Mineral Density Changes During Tx With Risperidone or Aripiprazole in Adolescents
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sriram Ramaswamy, M.D., Assistant Professor of Psychiatry, Creighton University
Other Study IDs: 06-14240
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Psychiatry
Keywords: bone mineral content; aripiprazole monotherapy; risperidone monotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 15 subjects who are taking aripiprazole monotherapy
- 2: 15 subjects who are taking Risperidone therapy
- 3: 30 healthy volunteers with an ethnicity, sex, and pubertal stage match of subjects taking aripiprazole monotherapy and Risperidone therapy

SUMMARY:
This study examines if the use of antipsychotic medications might contribute to an interruption in bone mineral development and/or a reduction in bone mineral content in adolescents.

DETAILED DESCRIPTION:
Studies have shown that some antipsychotic medications, including Risperdal, can increase prolactin levels in both adult and pediatric populations. Prolactin is a hormone made by the central nervous system. The main function of prolactin is to regulate lactation in females. However, having too much prolactin over time can interrupt bone mineral accrual and a decrease in bone density. Since peak bone mass is reached during adolescents, this is a key determinant of a lifetime risk of osteoporosis. On the other hand, there ahve been no reports of increased prolactin using Abilify. In fact, in adults Abilify has been shown to normalize or even lower prolactin levels. In this study, we will compare the amount of prolactin and bone mineral density of adolescents who take Risperdal or Abilify with bone mineral density of adolescents who do nto take antipsychotic medications. We will also compare the amount of prolactin and bone mineral density of adolescents who take Risperdal with those who take Abilify. This study will also help us to learn about the relationship between medications, prolactin levels, sex steroids, and bone formation markers in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 11 and 17 years
* Females and males on aripiprazole or risperidone monotherapy for minimum one year
* Within 10th and 90th percentile for height and weight

Exclusion Criteria:

* Pregnancy
* Chronic illness such as asthma, inflammatory bowel disease, rheumatoid disorders or cystic fibrosis, on chronic systemic steroid therapy for past 12 months
* Menstrual irregularities secondary to excessive physical activity
* History of anorexia nervosa and/or bulimia nervosa
* Subjects on hormonal contraception

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be recruited from psychiatry clinic and community resources
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
That compared to risperidone, pediatric aripiprazole therapy is not associated with hyperprolactinemia and reduced bone mineral content and/or altered bone metabolism | This is a 2-visit study

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Ramaswamy, M.D., Principal Investigator — Creighton University
Locations (1):
- Creighton Department of Psychiatry, Omaha, Nebraska, United States